CLINICAL TRIAL: NCT02946671
Title: Phase I Study of Pre-operative Combination Therapy With Mogamulizumab (Anti-CCR4) and Nivolumab (Anti-PD-1) Against Solid Cancer Patients
Brief Title: Study of Pre-operative Combination Therapy With Mogamulizumab and Nivolumab Against Solid Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Osaka University (Other)
Collaborators: Kyowa Kirin Co., Ltd. (Industry); Ono Pharmaceutical Co. Ltd (Industry); Clinical Study Support, Inc. (Unknown); Fiverings Co., Ltd. (Other)
Responsible Party: Principal Investigator, Hisashi Wada, Professor, Osaka University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KW0761-IIT-02
Record Dates: First submitted 2016-10-05; First posted 2016-10-27 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Gastric Cancer; Esophageal Cancer; Lung Cancer; Renal Cancer; Oral Cancer
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms; Lung Neoplasms; Kidney Neoplasms; Mouth Neoplasms | interventions — mogamulizumab; Nivolumab

ARMS (3):
- Cohort 1 (Experimental): KW-0761 (Mogamulizumab): 0.1 mg/kg, every week, 4 times ONO-4538 (Nivolumab): 3.0 mg/kg, every two weeks, 3 times
  Interventions: Biological: Mogamulizumab; Biological: Nivolumab
- Cohort 2 (Experimental): KW-0761 (Mogamulizumab): 0.3 mg/kg, every week, 4 times ONO-4538 (Nivolumab): 3.0 mg/kg, every two weeks, 3 times
  Interventions: Biological: Mogamulizumab; Biological: Nivolumab
- Cohort 3 (Experimental): KW-0761 (Mogamulizumab): 1.0 mg/kg, every week, 4 times ONO-4538 (Nivolumab): 3.0 mg/kg, every two weeks, 3 times
  Interventions: Biological: Mogamulizumab; Biological: Nivolumab

INTERVENTIONS:
Biological: Mogamulizumab — Mogamulizumab (0.1, 0.3 or 1.0 mg/kg) is administered.
  Other Names: KW-0761
Biological: Nivolumab — Nivolumab (3.0 mg/kg) is administered.
  Other Names: ONO-4538

SUMMARY:
To assess the safety of preoperative combination therapy with KW-0761 (anti-CCR4) and ONO-4538 (anti-PD-1).

To assess the behavior of immune cells in peripheral blood and tumor.

ELIGIBILITY:
Inclusion Criteria:

* Patients who enable to have standard operation
* Patients who refuse standard preoperative chemotherapy and are diagnosed with following cancers; gastric adenocarcinoma, esophageal squamous cell carcinoma, non-small-cell lung carcinoma, renal cell carcinoma or oral squamous cell carcinoma
* Patients with Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Patients with no serious disorder of major organs (born marrow, heart, lung, liver and kidney)
* Patients with written informed consent
* Patients who have measurable target lesion
* Patients who are enable to undergo biopsy for sampling tumor tissue

Exclusion Criteria:

* Known or previous autoimmune disease
* Known or suspected interstitial lung disease (ILD)
* Patients with history of serious anaphylaxis induced by antibody preparation
* Uncontrollable hypertension
* Uncontrollable endocrine disease
* Patients who have active inflammatory bowel disease or other serious GI chronic conditions associated with diarrhea
* Uncontrollable diabetes
* Prior therapy with sustained anticancer agents, radiotherapy or surgery for primary disease
* Pregnant or lactating females, female and male patients who cannot agree to practice the adequate birth control after the consent during the study
* Known or suspected infection or inflammatory disease
* Prior therapy with hematopoietic stem cell transplantation
* Known or suspected central nervous system (CNS) involvement

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-03; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events including intraoperative and postoperative complications | from first administration to 60 days after the final administration or to 30 days after the standard operation
  Confirm the toxicity profile, which is measured by the degree of grade and seriousness, duration, causality, classification, etc. of the adverse events.
Rate of Foxp3-positive patients in tumor by immunohistochemical analysis | from baseline until standard operation, an average of 7 weeks

SECONDARY OUTCOMES:
Objective tumor response rate according to RECIST v1.1 | from baseline to 6 weeks after the first administration
Rate of Treg decrease in peripheral blood mononuclear cell (PBMC) | from baseline to 60 days after the final administration or to 30 days after the standard operation

CONTACTS AND LOCATIONS:
Overall Officials: Hisashi Wada, M.D., Ph.D, Study Chair — Department of Clinical Research in Tumor Immunology, Graduate School of Medicine, Osaka University
Locations (1):
- Osaka University, Suita, Osaka, Japan

REFERENCES:
- [Derived] Jinushi K, Saito T, Kurose K, Suzuki S, Kojima T, Takahara T, Makino T, Ogawa T, Nishikawa H, Kakimi K, Iida S, Nakajima J, Doki Y, Oka M, Ueda R, Wada H. Phase I study on neoadjuvant combination immunotherapy with mogamulizumab and nivolumab for solid tumors. J Immunother Cancer. 2025 Apr 2;13(4):e010634. doi: 10.1136/jitc-2024-010634. PMID 40180420